CLINICAL TRIAL: NCT02724280
Title: Linked Color Imaging (LCI) System in the Identification of Normal Gastric Mucosa, Helicobacter Pylori Associated Gastritis and Gastric Atrophy
Brief Title: Linked Color Imaging to Differentiate H. Pylori Associated Gastritis and Gastric Atrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Collaborators: People's Hospital of Guangxi Zhuang Autonomous Region (Other); Shanghai 10th People's Hospital (Other); Second Affiliated Hospital of Soochow University (Other); Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 307-LCI-001
Record Dates: First submitted 2016-03-18; First posted 2016-03-31 (Estimated); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Gastritis; Helicobacter Pylori Associated Gastritis; Atrophic Gastritis
MeSH Terms: conditions — Gastritis; Gastritis, Atrophic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Active Comparator): Patients with indications for gastroduodenoscopy will be evaluated with WLE and then LCI.
  Interventions: Device: WLE and then LCI
- Group B (Placebo Comparator): Patients with indications for gastroduodenoscopy will be evaluated with LCI and then WLE.
  Interventions: Device: LCI and then WLE

INTERVENTIONS:
Device: WLE and then LCI — The gastric mucosa was evaluated with WLE and then LCI by two different endoscopists.
  Other Names: White light endoscopy (WLE) / linked color imaging (LCI)
  Arms: Group A
Device: LCI and then WLE — The gastric mucosa was evaluated with LCI and then WLE by two different endoscopists.
  Other Names: Linked color imaging (LCI) / White light endoscopy (WLE)
  Arms: Group B

SUMMARY:
H. pylori infection plays a very important role in gastric carcinogenesis, progressing from chronic gastritis through atrophic gastritis, intestinal metaplasia, dysplasia and finally cancer. It is difficult to diagnose H. pylori related gastritis and gastric atrophy on the basis of endoscopic findings. Histology is currently considered to be the gold standard for detecting H. pylori infection. The reliability of detecting H. pylori infection histologically depends on the site, number, and size of gastric biopsy specimens. The blind biopsy sampling of normal appearing mucosa has the risk of missing pathology and sampling errors. Most studies conclude that as well as on expertise in staining and visualizing the bacteria. Considerable error also occurs in identifying gastric atrophy using blind biopsy sampling, and neither the original nor the revised version of the Sydney system reliably identifies more than half the cases in patients with confirmed gastric atrophy.

DETAILED DESCRIPTION:
NBI is the most widely used system among several available image enhanced endoscopy systems. However, this technique has limitations such as dark imaging of distant lesions because of narrow-band illumination. Blue Laser Imaging (BLI) was developed to compensate for these inherent limitations of NBI. BLI uses narrow-band laser light combined with white light. This combination results in a bright image of the digestive mucosa, enabling the detailed visualization of both the microstructure and the microvasculature. However, BLI still is not able to obtain sufficient brightness for distant lesions. The newly developed Linked Color Imaging (LCI) system (FUJIFILM Co.) creates clear and bright endoscopic images by using short-wavelength narrow-band laser light combined with white laser light on the basis of BLI technology. This system can obtain bright endoscopic images even at a distant view because LCI has more intense white light than the short-wavelength narrow-band laser light. Short-wavelength narrow-band laser light enhances the vessels on the mucosal surface and the patterns of the mucosa, which means that BLI enables a clearer visualization of microvascular structures than does LCI. In contrast, LCI enhances differences in hue, in the red region of the spectrum, through digital processing. This makes red areas appear redder and white areas appear whiter. Thus, it is easier to recognize a slight difference in color of the mucosa. Therefore, LCI may facilitate the detection of H. pylori infection and gastric atrophy. Further studies are needed to confirm the utility of LCI.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old patients
* Who agree to participate in the study
* Patients with the indications for gastroduodenoscopy

Exclusion Criteria:

* Patients, who were receiving nonsteroidal anti-inflammatory drugs, pump inhibitors (PPI) or antibiotics in the last 3 weeks.
* Severe uncontrolled coagulopathy
* Prior history of gastric surgery.
* Pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Diagnosis rate of normal gastric mucosa, H. pylori associated gastritis and gastric atrophy | 6 months
  Number of patients with normal gastric mucosa, H. pylori associated gastritis and gastric atrophy will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Liu, M.D., Ph.D., Principal Investigator — Affiliated Hospital to Academy of Military Medical Sciences
Locations (1):
- Affiliated Hospital to Academy of Military Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Anagnostopoulos GK, Yao K, Kaye P, Fogden E, Fortun P, Shonde A, Foley S, Sunil S, Atherton JJ, Hawkey C, Ragunath K. High-resolution magnification endoscopy can reliably identify normal gastric mucosa, Helicobacter pylori-associated gastritis, and gastric atrophy. Endoscopy. 2007 Mar;39(3):202-7. doi: 10.1055/s-2006-945056. Epub 2007 Feb 1. PMID 17273960
- [Result] Yao K, Anagnostopoulos GK, Ragunath K. Magnifying endoscopy for diagnosing and delineating early gastric cancer. Endoscopy. 2009 May;41(5):462-7. doi: 10.1055/s-0029-1214594. Epub 2009 May 5. PMID 19418401